CLINICAL TRIAL: NCT00632749
Title: An Open Phase I/IIa Trial to Investigate the Maximum Tolerated Dose, Safety, Efficacy and Pharmacokinetics of BI 811283 in Combination With Cytarabine in Patients With Previously Untreated Acute Myeloid Leukaemia Ineligible for Intensive Treatment
Brief Title: BI 811283 in Combination With Cytarabine in Previously Untreated AML Ineligible for Intensive Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1247.3; 2007-005684-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

ARMS (2):
- Schedule A (Experimental): BI 811283 on days 1 and 15 in combination with Cytarabine 20 mg twice daily on Days 1-10
  Interventions: Drug: BI 811283 (d 1 and 15); Drug: Cytarabine
- Schedule B (Experimental): BI 811283 on Day 1 in combination with Cytarabine 20 mg twice daily on Days 1-10
  Interventions: Drug: Cytarabine; Drug: BI 811283 (d1)

INTERVENTIONS:
Drug: BI 811283 (d 1 and 15) — BI 811283 (24 hours i.v.c.i.) on day 1 and 15 of a 4-week treatment cycle
  Arms: Schedule A
Drug: Cytarabine — Cytarabine 2 x 20 mg/d s.c. on days 1-10 of a 4-week treatment cycle
  Arms: Schedule B
Drug: BI 811283 (d1) — BI 811283 (24 hours i.v.c.i.) on day 1 of a 4-week treatment cycle
  Arms: Schedule B
Drug: Cytarabine — Cytarabine 2 x 20 mg/d s.c. on days 1-10 of a 4-week treatment cycle
  Arms: Schedule A

SUMMARY:
Investigation of maximum tolerated dose, safety, efficacy and pharmcokinetics of BI 811283 in combination with cytarabine (LD-Ara-C) in previously untreated acute myeloid leukaemia (AML) patients

ELIGIBILITY:
Inclusion criteria:

* Male or female adult with previously untreated acute myeloid leukaemia (AML)
* Confirmed diagnosis of AML according to the WHO definition (except for acute promyelocytic leukaemia, APL)
* Patient is considered ineligible for intensive treatment
* Patient is eligible for low-dose cytarabine (LD-Ara-C) treatment
* Life expectancy > 3 months
* Eastern co-operative oncology group (ECOG, R01-0787) performance score <=2 at screening
* Signed written informed consent consistent with international conference on harmonisation good clinical practice (ICH-GCP) and local legislation

Exclusion criteria:

* Patient with APL (AML subtype M3 according to the French-American-British (FAB) classification).
* Relapsed or treatment refractory AML.
* Hypersensitivity to one of the trial drugs or the excipients.
* Other malignancy requiring treatment.
* Known central nervous system involvement.
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (ULN).
* INR > 1.5 x ULN for subjects not on therapeutic vitamin K antagonists (phenprocoumon, warfarin).
* Bilirubin greater than 1.5 mg/dl.
* Serum creatinine greater than 2.0 mg/dl.
* LVEF (Left ventricular ejection fraction) < 50% in echocardiography or clinical congestive heart failure New York Heart Association (NYHA) grade III or IV.
* Concomitant intercurrent illness, which would compromise the evaluation of efficacy or safety of the trial drug, e.g. active severe infection, unstable angina pectoris or cardiac arrhythmia.
* Psychiatric illness or social situation that would limit compliance with trial requirements.
* Concomitant therapy, which is considered relevant for the evaluation of the efficacy or safety of the trial drug (i.e. other chemo- or immunotherapy, see also section 4.2.2).
* Contraindications for cytarabine treatment according to the summary of product characteristics (SPC).
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception during the trial (hormonal contraception, intrauterine device, condom with spermicide, etc.).
* Pregnant or nursing female patients.
* Patient unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Germany (7):
  - 1247.3.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 1247.3.49005 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1247.3.49004 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1247.3.49006 Boehringer Ingelheim Investigational Site, Hamburg
  - 1247.3.49003 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1247.3.49002 Boehringer Ingelheim Investigational Site, Münster
  - 1247.3.49001 Boehringer Ingelheim Investigational Site, Ulm

REFERENCES:
- [Derived] Dohner H, Muller-Tidow C, Lubbert M, Fiedler W, Kramer A, Westermann J, Bug G, Schlenk RF, Krug U, Goeldner RG, Hilbert J, Taube T, Ottmann OG. A phase I trial investigating the Aurora B kinase inhibitor BI 811283 in combination with cytarabine in patients with acute myeloid leukaemia. Br J Haematol. 2019 May;185(3):583-587. doi: 10.1111/bjh.15563. Epub 2018 Nov 19. No abstract available. PMID 30450591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 participants were entered, and 64 were treated with the study treatment
Groups:
- 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A: 5 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A: 15 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A: 30 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A: 60 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A: 100 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A: 120 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 5 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 40 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 80 mg BI 811283+ 20 mg Cytarabine - Treatment Schedule B: 80 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 160 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 240 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 300 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 360 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 420 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
Period: Overall Study
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283+ 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Started | 4 | 5 | 3 | 4 | 7 | 8 | 5 | 4 | 5 | 3 | 7 | 4 | 3 | 6
Treated | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
Not Treated | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 3 | 4 | 7 | 8 | 5 | 4 | 5 | 3 | 7 | 4 | 3 | 6
Not completed — Progressive disease | 3 | 2 | 2 | 2 | 4 | 4 | 3 | 2 | 3 | 2 | 4 | 3 | 2 | 4
Not completed — Other Adverse event | 1 | 1 | 1 | 1 | 2 | 4 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Refuse to continue medication | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Reason other than those specified above | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 68 participants were randomised, and 64 were treated with the study treatment hence the number of participants differs from the number of participants that started in the participant flow.
Groups:
- 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B: 80 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | Total
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (5.8) | 71.3 (2.5) | 79.3 (8.4) | 77.5 (4.0) | 67.4 (9.3) | 72.3 (5.1) | 74.3 (4.1) | 73.5 (6.6) | 79.0 (4.4) | 78.3 (4.0) | 72.3 (4.4) | 69.5 (11.8) | 63.3 (5.1) | 63.3 (5.6) | 72.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 4 | 3 | 1 | 3 | 2 | 2 | 2 | 2 | 0 | 2 | 30
  Male | 1 | 1 | 1 | 2 | 3 | 4 | 3 | 1 | 3 | 1 | 5 | 2 | 3 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of 2 Schedules of BI 811283 in Combination With Cytarabine.
Description: The MTD was defined as the highest dose at which 6 patients were treated and less than 2 patients who experienced a dose limiting toxicities (DLT) within the first cycle of treatment.The MTD was defined based on safety data from the first cycle only.
  It was determined using a standard "3 + 3 design with de-escalation".
Time Frame: up to 28 days of treatment
Population: Treated set (TS): All patients who received at least one single dose of trial medication (BI 811283 or cytarabine) were considered.
Measure: Number; unit: mg
Groups:
- Treatment Schedule A: Subjects received BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle).
  BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection).
  The starting dose for BI 811283 was 5 mg, with dose levels of 5, 15, 30, 60, 100 and 120 mg used in Schedule A.
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- Treatment Schedule B: Subjects received BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle).
  BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection).
  The starting dose for BI 811283 was 5 mg, with dose levels of 5, 40, 80, 160, 240, 300, 360 and 420 mg being used in Schedule B.
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
Arm/Group | Treatment Schedule A | Treatment Schedule B
Number analyzed (Participants) | 28 | 36
mg | 100 | NA — Due to the early termination of the study for strategic reasons, the MTD was not reached in Schedule B

2. Secondary Outcome: Response (Complete Remission [CR], Complete Remission With Incomplete Blood Count Recovery [CRi])
Description: Response to treatment was evaluated according to the following criteria (modified from the National Cancer Institute/Cancer and Leukemia Group B criteria:
  The best overall response was defined as the best overall response recorded during the time period from the start of the treatment until the end of the treatment period, progression or death (whichever was earlier). Possible categories for best overall response were CR, CRi, Partial remission (PR), no change (NC), Progressive disease (PD) and no assessment.
  * Complete remission (CR): morphologically leukaemia free state (i.e. bone marrow with < 5% blasts by morphologic criteria and no Auer rods, no evidence of extramedullary leukaemia) and absolute neutrophil count ≥ 1,000/μL and platelets > 100,000/μL.
  * Complete remission with incomplete blood count recovery ("incomplete" CR, CRi).All of the above criteria for CR had to be met, except that neutrophils < 1,000/μL or platelets < 100,000/μL in the blood.
Time Frame: Data collected up to cut-off date 20Oct2011, Up to 1239 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
participants
  CR | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
  CRi | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Incidence and Intensity of AEs Graded According to CTCAE (Version 3.0)
Description: The severity and timing of AEs indicates how well the treatment regimen was tolerated.
  Toxicities were evaluated using the common terminology criteria for adverse events (CTCAE) grading scheme.
Time Frame: Data from first treatment administration until cut-off date of 20 October 2011; up to 1239 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
participants
  CTCAE Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CTCAE Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CTCAE Grade 3 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0
  CTCAE Grade 4 | 0 | 2 | 2 | 2 | 4 | 3 | 1 | 2 | 3 | 1 | 3 | 1 | 2 | 2
  CTCAE Grade 5 | 3 | 0 | 0 | 1 | 2 | 4 | 2 | 2 | 2 | 1 | 2 | 2 | 1 | 4

4. Secondary Outcome: Incidence of Dose Limiting Toxicity (DLT)
Description: Number of participants with DLT in the first cycle (28 days) for the determination of the maximum tolerated dose (MTD)
Time Frame: up to 28 days of treatment
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
participants | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0

5. Secondary Outcome: Partial Remission
Description: Response to treatment was evaluated according to the following criteria (modified from the National Cancer Institute/Cancer and Leukemia Group B criteria; The best overall response was defined as the best overall response recorded during the time period from the start of the treatment until the end of the treatment period, progression or death (whichever was earlier). Possible categories for best overall response were CR, CRi, Partial remission (PR), no change (NC), Progressive disease (PD) and no assessment.
  Partial remission (PR). All of the criteria for CR had to be met, except that the bone marrow had to contain ≥ 5% but less than 25% blasts (or ≤ 50% of initial blast count), or < 5% blasts in the presence of Auer rods or abnormal morphology.
Time Frame: Data collected up to cut-off date 20 Oct 2011, Up to 1239 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the duration of time from randomisation to time of treatment failure (i.e. PD), relapse from CR, or death from any cause, whichever came first.
Time Frame: Data collected up to cut-off date 20 Oct 2011, Up to 1239 days
Population: Treated set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
days | 35.0 (15.6) | 122.3 (120.0) | 32.0 (1.0) | 117.5 (102.4) | 60.4 (52.6) | 62.0 (54.1) | 209.0 (315.8) | 65.0 (41.5) | 168.8 (219.3) | 62.7 (53.9) | 138.7 (183.2) | 48.5 (36.9) | 174.0 (67.2) | 30.0 (7.3)

7. Secondary Outcome: Relapse Free Survival
Description: Relapse-free survival was defined only for patients who achieved CR/CRi and was measured from the date of attaining CR/CRi until the date of recurrence or death from any cause, whichever occurred first.
  Number of patients having relapse free survival are presented.
Time Frame: Data collected up to cut-off date 20 Oct 2011, Up to 1239 days
Population: Treated set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: participants
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0
participants |  |  |  | 1 |  | 1 | 1 |  | 1 | 1 | 1 |  | 2 |

8. Secondary Outcome: Remission Duration
Description: Remission duration analysis was defined only for patients who achieved CR, and was measured from the date of attaining CR until the date of disease recurrence (relapse). For patients who died without report of relapse, remission duration was censored on the date of death, regardless of the cause.
Time Frame: Data collected up to cut-off date 20 Oct 2011, Up to 1239 days
Population: Treated set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Deviation); unit: days
Groups:
- 240 mg BI 811283+ 20 mg Cytarabine - Treatment Schedule B: 240 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283+ 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
days |  |  |  | 263.0 (NA) — As only one participant is analyzed, SD is not calculable |  | 28.0 (NA) — As only one participant is analyzed, SD is not calculable | 337.0 (NA) — As only one participant is analyzed, SD is not calculable |  | 455.0 (NA) — As only one participant is analyzed, SD is not calculable |  | 128.0 (NA) — As only one participant is analyzed, SD is not calculable |  | 15.0 (NA) — As only one participant is analyzed, SD is not calculable |

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined for all patients that entered the trial, and measured from the date of randomization until death from any cause.
Time Frame: Data collected up to cut-off date 20 Oct 2011, Up to 1239 days
Population: Treated set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 4 | 3 | 6
days | 122.8 (166.2) | 212.0 (55.1) | 71.3 (40.5) | 236.8 (225.5) | 148.7 (125.5) | 86.6 (58.1) | 236.8 (322.9) | 137.3 (121.7) | 198.2 (260.1) | 339.7 (364.8) | 175.7 (175.4) | 73.0 (31.3) | 294.7 (101.5) | 48.7 (17.9)

10. Secondary Outcome: Cmax (Maximum Measured Concentration of BI 811283 in Plasma)
Description: Cmax (maximum measured concentration of BI 811283 in plasma) during Cycle 1
Time Frame: -0.05 hours before and 1:00, 4:00, 6:00, 24:00, 25:00, 26:00, 28:00, 32:00, 36:00, 48:00 hours after administration of BI 811283
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- 30 mg BI 811283 + 20 mg Cytarabine- Treatment Schedule A: 30 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
- 120mg (BI 811283+ Cytarabine)- Treatment Schedule A: 120 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment Schedule A: BI 811283 on Days 1 + 15 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine- Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120mg (BI 811283+ Cytarabine)- Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 3 | 3 | 6
nmol/L | 8.03 (32.3) | 64.10 (686.0) | 104.00 (321.0) | 153.00 (108.0) | 214.00 (38.8) | 272.00 (30.0) | 7.06 (10.0) | 66.10 (85.3) | 139.00 (33.8) | 499.00 (101.0) | 445.00 (71.0) | 631.00 (31.0) | 528.00 (40.5) | 1130.00 (53.3)

11. Secondary Outcome: AUC(0-inf) (Area Under the Concentration-time Curve of BI 811283 in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC(0-inf) (area under the concentration-time curve of BI 811283 in plasma over the time interval from 0 extrapolated to infinity) during Cycle 1
Time Frame: as for outcome 10
Population: Treated set (Only patients with observed cases (OC) values were analysed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol·h/L
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 2 | 3 | 6 | 7 | 4 | 4 | 5 | 3 | 7 | 3 | 3 | 6
nmol·h/L | 177 (28.2) | 985 (311.0) | 1000 (40.7) | 2790 (130) | 4400 (62.9) | 5620 (27.9) | 192 (47.7) | 1490 (98.1) | 2840 (29.6) | 8870 (59.9) | 9770 (63.0) | 14100 (32.6) | 12800 (64.3) | 23200 (57.9)

12. Secondary Outcome: AUC0-tz (Area Under the Concentration-time Curve of BI 811283 in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: AUC0-tz (area under the concentration-time curve of BI 811283 in plasma over the time interval from 0 to the time of the last quantifiable data point) during Cycle 1
Time Frame: as for outcome 10
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol·h/L
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 3 | 3 | 6
nmol·h/L | 169 (30.5) | 939 (328) | 2010 (207) | 2350 (105) | 2810 (135) | 5340 (27.2) | 156 (17.5) | 1450 (97.3) | 2730 (29.1) | 8680 (60.4) | 9260 (63.6) | 13700 (31.7) | 12100 (63.1) | 21700 (55.2)

13. Secondary Outcome: Cmax,ss (Maximum Measured Concentration of BI 811283 in Plasma at Steady State)
Description: Cmax (maximum measured concentration of BI 811283 in plasma at steady state) during Cycle 1
Time Frame: as for outcome 10
Population: Treated set (Only patients with observed cases (OC) values were analysed). Steady state analyses is not applicable for Treatment Schedule B, since pharmacokinetic analyses was performed after a single dose for Treatment Schedule B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 7
nmol/L | 8.02 (4.59) | 24.7 (18.5) | 43.3 (5.58) | 141 (52.2) | 213 (96.1) | 229 (67.9)

14. Secondary Outcome: AUC (0-inf, ss)(Area Under the Concentration-time Curve of BI 811283 in Plasma Over the Time Interval From 0 Extrapolated to Infinity) at Steady State
Description: AUC (0-inf, ss)(area under the concentration-time curve of BI 811283 in plasma over the time interval from 0 extrapolated to infinity) at steady state during Cycle 1
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol·h/L
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 6 | 7
nmol·h/L | 188 (12.7) | 615 (15.3) | NA (NA) — Not calculated as estimates of summary statistical values are not considered reliable if data from fewer than 2/3 of tested subjects are available, according to Boehringer-Ingelheim Clinical PK SOP | 4460 (41.8) | 5140 (105.0) | 4750 (58.1)

15. Secondary Outcome: AUC (0-tz,ss) (Area Under the Concentration-time Curve of BI 811283 in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point) at Steady State
Description: AUC (0-tz,ss) (area under the concentration-time curve of BI 811283 in plasma over the time interval from 0 to the time of the last quantifiable data point) at steady state during Cycle 1
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol·h/L
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 7
nmol·h/L | 183 (14.3) | 597 (15.0) | 1620 (58.2) | 4330 (40.5) | 4340 (83.6) | 4820 (55.6)

16. Secondary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration of BI 811283 in Plasma)
Description: tmax (time from dosing to maximum measured concentration of BI 811283 in plasma) during Cycle 1
Time Frame: as for outcome 10
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Median (Full Range); unit: hours
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 7 | 7 | 4 | 4 | 5 | 3 | 7 | 3 | 3 | 6
hours | 24.0 [6.0 to 24.1] | 26.0 [6.0 to 48.0] | 25.0 [24.0 to 32.0] | 22.7 [6.0 to 24.1] | 6.0 [4.1 to 24.3] | 23.6 [5.9 to 24.5] | 23.9 [4.0 to 24.2] | 6.0 [6.0 to 6.0] | 24.1 [6.0 to 26.8] | 24.9 [23.6 to 32.0] | 6.0 [6.0 to 25.0] | 23.9 [23.9 to 24.1] | 5.9 [4.8 to 6.0] | 14.8 [3.9 to 26.1]

17. Secondary Outcome: Tmax,ss (Time From Dosing to Maximum Measured Concentration of BI 811283 in Plasma at Steady State)
Description: tmax,ss (time from dosing to maximum measured concentration of BI 811283 in plasma at steady state) during Cycle 1
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 7
hours | 23.9 [4.1 to 23.9] | 24.0 [4.0 to 24.0] | 6.0 [4.0 to 24.0] | 6.0 [4.1 to 24.0] | 6.0 [5.9 to 23.5] | 6.0 [4.0 to 23.8]

18. Secondary Outcome: Cmax (Maximum Measured Concentration of Cytarabine in Plasma)
Description: Cmax of Cytarabine after a 20 mg Subcutaneous Dose on the First Day of BI 811283
Time Frame: -0.05 hours before and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 hours after administration of Cytarabine
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 6 | 7 | 4 | 3 | 5 | 3 | 7 | 3 | 3 | 6
ng/mL | 53.2 (65.4) | 72.6 (31.0) | 49.0 (80.6) | 64.9 (49.5) | 61.9 (57.3) | 46.0 (54.1) | 46.3 (31.8) | 49.8 (58.1) | 55.0 (16.5) | 65.1 (44.5) | 49.4 (58.9) | 48.6 (88.4) | 49.0 (77.0) | 68.7 (33.1)

19. Secondary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration of Cytarabine in Plasma)
Description: Tmax of Cytarabine after a 20 mg Subcutaneous Dose on the First Day of BI 811283
Time Frame: -0.05 hours before and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 hours after administration of Cytarabine
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Median (Full Range); unit: hours
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 6 | 7 | 4 | 3 | 5 | 3 | 7 | 3 | 3 | 6
hours | 0.50 [0.50 to 1.0] | 0.50 [0.50 to 1.0] | 0.92 [0.50 to 1.0] | 0.83 [0.50 to 1.4] | 0.48 [0.42 to 0.53] | 0.55 [0.50 to 1.5] | 0.50 [0.40 to 0.70] | 0.50 [0.50 to 0.50] | 0.58 [0.47 to 1.0] | 0.50 [0.43 to 0.67] | 0.50 [0.45 to 1.0] | 0.50 [0.47 to 0.50] | 0.48 [0.48 to 1.0] | 0.49 [0.48 to 0.57]

20. Secondary Outcome: AUC (0-inf) (Area Under the Concentration-time Curve of Cytarabine in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC (0-inf) of Cytarabine after a 20 mg Subcutaneous Dose on the First Day of BI 811283
Time Frame: -0.05 hours before and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 hours after administration of Cytarabine
Population: Treated set (Only patients with observed cases (OC) values were analysed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 4 | 5 | 4 | 2 | 3 | 3 | 7 | 3 | 2 | 5
ng·h/mL | 104 (31.4) | 122 (6.89) | 102 (31.5) | 85.4 (35.3) | 65.9 (42.5) | 68.1 (41.4) | 62.0 (24.1) | NA (NA) — Not calculated as estimates of summary statistical values are not considered reliable if data from fewer than 2/3 of tested subjects are available, according to Boehringer-Ingelheim Clinical PK SOP | NA (NA) — Not calculated as estimates of summary statistical values are not considered reliable if data from fewer than 2/3 of tested subjects are available, according to Boehringer-Ingelheim Clinical PK SOP | 71.2 (20.7) | 72.7 (23.6) | 75.5 (27.2) | 76.9 (19.5) | 76.8 (42.6)

21. Secondary Outcome: AUC (0-tz) (Area Under the Concentration-time Curve of Cytarabine in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: AUC (0-tz) of Cytarabine after a 20 mg Subcutaneous Dose on the First Day of BI 811283
Time Frame: -0.05 hours before and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 hours after administration of Cytarabine
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/L
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 6 | 7 | 4 | 3 | 5 | 3 | 7 | 3 | 3 | 6
ng·h/L | 45.0 (156.0) | 66.9 (73.8) | 66.8 (57.6) | 71.8 (26.4) | 46.6 (51.2) | 42.3 (64.3) | 45.9 (20.0) | 33.9 (245.0) | 57.0 (18.2) | 60.2 (30.4) | 52.5 (38.8) | 52.1 (42.1) | 41.3 (87.2) | 51.6 (38.1)

22. Secondary Outcome: Pharmacodynamic Monitoring
Description: Pharmacodynamic monitoring: drug effect on leukaemia cells (e.g. polyploidy, histone H3 phosphorylation, morphologic changes).
  An evaluation of this secondary endpoint is not possible due to missing samples / samples of poor quality of the provided material.
Time Frame: On Day 5, i.e. 72 hours after the end of the first BI 811283 infusion, and on Day 28 in the first cycle only
Population: Treated set
Groups:
- 80 mg BI 811283 +20 mg Cytarabine - Treatment Schedule B: 80 mg of BI 811283 (preconcentrate for infusion after dilution) in combination with cytarabine (solution for injection);
  Treatment schedule B: BI 811283 on Day 1 in combination with cytarabine 20 mg twice daily on Days 1-10 (28-day cycle);
  BI 811283: 24-hour continuous intravenous infusion Cytarabine: subcutaneous injection
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 +20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Pharmacokinetics of Cytarabine After a Single Dose and at Steady State When Given Alone
Description: The study protocol originally included a phase II part with a treatment arm in which Cytarabine was given alone, however the sponsor discontinued the clinical development of BI 811283, therefore the protocol was amended and the reference therapy arm was removed from the study protocol" -> (Protocol Amendment 5, version 19 -May-2010, approved 28-Jun-2010).
  Since there was never a treatment arm in which Cytarabine was given alone; hence pharmacokinetics are not calculated.
Time Frame: -0.05, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00 hours
Population: Treated set
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Data from first treatment administration until cut-off date of 20 October 2011; up to 1239 days
Arm/Group | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 3/3 | 4/4 | 6/7 | 6/7 | 4/4 | 3/4 | 5/5 | 3/3 | 7/7 | 3/4 | 3/3 | 5/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 4/4 | 7/7 | 7/7 | 4/4 | 4/4 | 5/5 | 3/3 | 6/7 | 4/4 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=4) | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=3) | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=3) | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=4) | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=7) | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=7) | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=4) | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=4) | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=5) | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=3) | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=7) | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=4) | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=3) | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=6)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 3 | 1 | 1 | 1 | 2 | 2 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=4) | 15 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=3) | 30 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=3) | 60 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=4) | 100 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=7) | 120 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule A (N=7) | 5 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=4) | 40 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=4) | 80 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=5) | 160 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=3) | 240 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=7) | 300 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=4) | 360 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=3) | 420 mg BI 811283 + 20 mg Cytarabine - Treatment Schedule B (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 5 | 5 | 1 | 2 | 1 | 3 | 3 | 1 | 3 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 4 | 5 | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 3 | 3 | 2 | 2 | 2 | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid bleeding (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 1 | 1 | 3 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 3 | 4 | 1 | 1 | 3 | 2 | 1 | 3 | 3 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 4 | 3 | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 1 | 3 | 2 | 1 | 2 | 1 | 3 | 4 | 2 | 1 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3
Inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0
Pain (General disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 1 | 3 | 2 | 4 | 1 | 2 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic vein occlusion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Basophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood cholinesterase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 5 | 4 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 4 | 2 | 2 | 0 | 0 | 0 | 4 | 1 | 2 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mean cell haemoglobin concentration increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mean cell volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Prothrombin time shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
pH urine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 4 | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 3 | 2 | 1 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Spinal haematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Catatonia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Illusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 2 | 3 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 4 | 1 | 2 | 1 | 3 | 5 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bedridden (Social circumstances) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheterisation venous (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 0 | 2 | 1 | 2 | 2 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.